CLINICAL TRIAL: NCT00273663
Title: The Effects of Transcranial Electrical Stimulation (TCES) on Cerebral Blood Flow (CBF) With Xenon Under Computerized Tomography (Xe/CT)
Brief Title: Transcranial Electrical Stimulation (TCES) / Cerebral Blood Flow (CBF) / Xenon Under Computerized Tomography (Xe/CT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9376-03; 2003-038
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2007-06

CONDITIONS: Healthy Volunteers
Keywords: cerebral blood flow; electrical stimulation; Computed Tomography Scanner, X-Ray; Brain Mapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: TCES

SUMMARY:
Direct stimulation of the cerebral cortex induces an increase in cerebral blood flow. Although this information is known, it has never been documented during Transcranial Cerebral Electrical Stimulation (TCES), which is a non invasive technique. It is used to modulate the opiate endogenous system, mainly in opioid users but no cerebral blood flow mapping of the anatomic regions involved in this modulation of the opiate system under electrical stimulation has been performed in functional Computerized Tomography.

DETAILED DESCRIPTION:
* Principal Objective : To compare the increase in mean cerebral blood flow in a group of defined zones (the thalamus, anterior cingulate gyrus, the insula, periacqueductal region of the brain stem,the frontal lobes, the striatum and limbic system) in healthy volunteers stimulated or not stimulated by TCES.
* Secondary Objective : Description of cerebral blood flow variations in the different zones in order to map electrostimulated areas.
* Study design : An experimental, randomized, double-blind, single-centre trial with 2 groups, a study group (stimulated by TCES) and a control group (not stimulated).
* Inclusion criteria : Participants free of any known neurological or psychiatric disorder; participants not under treatment particularly with opioids, analgesics or medication containing codeine or morphine for at least a month; participants aged between 18 and 65 having signed a written informed consent ; participants having accepted to be registered on the national eligibility list for subjects participating in a trial without direct individual benefit, and covered by an insurance policy.
* Exclusion criteria : Participation in two different study trials without direct individual benefit at the same time. Contraindications to Computerized Tomography. Subjects diagnosed clinically with a Neurological or Psychiatric disorder; Subjects who have been under analgesics or morphine agonists for less than a month; Pregnant or breastfeeding mothers and women without an adequate contraception. Drug addicts or persons under tutelage.
* Study plan: Study group: Xe/CT and transcranial electrostimulation / Control group : Xe/CT
* Principal Criterion of Judgement: difference in mean cerebral blood flow between the study group(stimulated) and the control group (not stimulated).
* Secondary Criteria of Judgement : Difference in mean cerebral blood flow region per region (thalamus, anterior cingulate gyrus, insula, periacqueductal region of the brain stem, the frontal lobes, the striatum and limbic system).
* Number of subjects : 40
* Duration of subject participation in study : 2 H 30

ELIGIBILITY:
Inclusion Criteria:

* Participants free of any known neurological or psychiatric disorder
* participants not under treatment particularly with opioids, analgesics or medication containing codeine or morphine for at least a month
* 18 and 65
* informed consent signed

Exclusion Criteria:

* Contraindications to Computerized Tomography
* Subjects diagnosed clinically with a Neurological or Psychiatric disorder
* Subjects who have been under analgesics or morphine agonists for less than a month
* Pregnant or breastfeeding mothers and women without an adequate contraception
* Drug addicts
* persons under tutelage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
difference in mean cerebral blood flow between the study group(TCES stimulated) and the control group (TCES not stimulated).

SECONDARY OUTCOMES:
Difference in mean cerebral blood flow zone per zone (thalamus, anterior cingulate gyrus, insula, periacqueductal region of the brain stem, the frontal lobes, the striatum and limbic system).

CONTACTS AND LOCATIONS:
Overall Officials: Patrice MENEGON, MD, Principal Investigator — University Hospital, Bordeaux; Rodolphe THIEBAUT, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- Service de Neuro-radiologie, hôpital Pellegrin, Bordeaux, France

REFERENCES:
- [Derived] Gense de Beaufort D, Sesay M, Stinus L, Thiebaut R, Auriacombe M, Dousset V. Cerebral blood flow modulation by transcutaneous cranial electrical stimulation with Limoge's current. J Neuroradiol. 2012 Jul;39(3):167-75. doi: 10.1016/j.neurad.2011.06.001. Epub 2011 Aug 10. PMID 21835468